CLINICAL TRIAL: NCT01629862
Title: Vascular Impairment in Type II Diabetes Mellitus With Co-morbid Obstructive Sleep Apnea.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanjay R Patel (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Sanjay R Patel, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8354706
Record Dates: First submitted 2012-05-08; First posted 2012-06-28 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea, Obstructive; Diabetes Mellitus
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active CPAP (Active Comparator): Therapeutic continuous positive airway pressure (CPAP).
  Interventions: Device: Continuous positive airway pressure
- Sham CPAP (Placebo Comparator): Sham (non-therapeutic) continuous positive airway pressure.
  Interventions: Device: Sham continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — CPAP at therapeutic pressure; ResMed S9 device in fixed pressure mode (Sydney, Australia).
  Arms: Active CPAP
Device: Sham continuous positive airway pressure — CPAP at non-therapeutic pressure; ResMed S9 device using a ResMed sham mask (Sydney, Australia).
  Arms: Sham CPAP

SUMMARY:
The investigators will examine the possible synergistic effects of obstructive sleep apnea (OSA) and type II diabetes mellitus (DM) on vascular functioning by performing a two-part investigation:

* A cross-sectional study comparing subjects with OSA+DM, OSA only, DM only, and healthy controls.
* A three-month randomized placebo-controlled trial of continuous positive airway pressure (CPAP) in subjects with OSA+DM.

ELIGIBILITY:
Inclusion Criteria:

* OSA subjects: apnea-hypopnea index >=10 and <100
* DM subjects: clinical diagnosis of DM and glycated hemoglobin < 8.0%

Exclusion Criteria:

* Hematocrit < 32
* Pregnancy
* Infectious/collagen vascular/hepatic or renal/cardiopulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aristidis Veves, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Sanjay R Patel, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] Bakker JP, Baltzis D, Tecilazich F, Chan RH, Manning WJ, Neilan TG, Wallace ML, Hudson M, Malhotra A, Patel SR, Veves A. The Effect of Continuous Positive Airway Pressure on Vascular Function and Cardiac Structure in Diabetes and Sleep Apnea. A Randomized Controlled Trial. Ann Am Thorac Soc. 2020 Apr;17(4):474-483. doi: 10.1513/AnnalsATS.201905-378OC. PMID 31922899

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active CPAP | Sham CPAP
Started | 28 | 25
Completed | 26 | 23
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CPAP | Sham CPAP | Total
Number analyzed (Participants) | 28 | 25 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 14 | 14 | 28
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Brachial Artery Flow-mediated Dilation (FMD).
Description: Brachial artery flow-mediated dilation is measured as the percent change in brachial artery diameter post-occlusion relative to pre-occlusion. The change in brachial artery flow mediated dilation is the difference in this percent change at 3-months compared to baseline.
Time Frame: 3 months (compared to baseline)
Measure: Mean (Standard Deviation); unit: percentage of brachial artery diameter
Arm/Group | Active CPAP | Sham CPAP
Number analyzed (Participants) | 26 | 23
percentage of brachial artery diameter | 2.26 (3.80) | 1.59 (4.85)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Regular investigator assessment of adverse events (at each visit and follow-up phone call)
Arm/Group | Active CPAP | Sham CPAP
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/28 | 1/25
Other Adverse Events (participants affected / at risk) | 1/28 | 5/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=28) | Sham CPAP (N=25)
Spinal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary artery bypass surgery (Cardiac disorders) | 0 (0) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — After planned surgery, requiring reoperation
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active CPAP (N=28) | Sham CPAP (N=25)
Asthenia (Psychiatric disorders) | 0 (0) | 1 (1) — Felt psychogenic etiology after clinical evaluation
Broken arm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
IV infiltration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vasovagal reaction (Cardiac disorders) | 0 (0) | 1 (1) — Following blood draw. Cause unknown; similar episodes reported over a matter of weeks.
Hit by falling snow (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Persistent bleeding at skin biopsy site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT01629862/SAP_000.pdf
  • Study Protocol (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT01629862/Prot_001.pdf